CLINICAL TRIAL: NCT04719676
Title: Comparison of Core Strength Training Using Stable Versus Unstable Surfaces On Strength, Flexibility, Balance, Coordination and Speed in Gym Members
Brief Title: Comparison of Core Strength Training Using Stable Versus Unstable Surfaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00718 Raeed Mufti
Record Dates: First submitted 2020-11-15; First posted 2021-01-22 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Sports Physical Therapy
Keywords: Core Strength Training; Flexibility; Balance; Coordination; Speed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core strength training using unstable surface (Experimental): The experimental group will use Core strength training using unstable surface
  Interventions: Other: Core strength training using unstable surface
- The stable surface would be gym floor. (Active Comparator): The control group will use stable surface.
  Interventions: Other: The stable surface would be gym floor.

INTERVENTIONS:
Other: Core strength training using unstable surface — Training would include "big 3" exercises as described by McGill. These include the curl-up, side bridge, and quadruped position on unstable surface
  Arms: Core strength training using unstable surface
Other: The stable surface would be gym floor. — Training would include "big 3" exercises as described by McGill. These include the curl-up, side bridge, and quadruped position on stable gym Floor
  Arms: The stable surface would be gym floor.

SUMMARY:
This study will address the scarcity of research and the variations in recommendations regarding core strengthening and stability programs. As physical fitness is a major concern of individuals and mostly people refer gym for fitness enhancement, this study will thus provide a guideline for effective core strength training program

DETAILED DESCRIPTION:
Male clients, aged 19 to 44 years, coming to the gym for strength training will be purposively selected based on the inclusion criteria and then randomly assigned into two groups. They will undergo a series of pre-intervention tests that would assess their strength using Bourbon TMS and standing long jump tests; flexibility using stand and reach test; balance using Y balance test; coordination using jumping sideways test and speed using 20-m sprint test. After initial assessment, they will be advised and demonstrated for curl-up, side-bridging and quadrupled exercises. The experimental group will perform these exercises on Thera-Band© Exercise Ball while the control group will perform the same exercises on gym floor. The clients will have sessions on preferably the first day and 4th day of the week but is subject to their attendance at the gym. There will be interval assessments at 2nd and 4th week based on the tests mentioned above to record changes at these intervals. After 6 weeks of bi-weekly sessions, the clients will undergo post-intervention tests that will be the same as pre-intervention tests.

ELIGIBILITY:
Inclusion Criteria:

* Male clients
* Male adults with age 19-44 years
* Regular gym attendance with at least two gym workout session per week

Exclusion Criteria:

* Recent history of injury or illness
* Clients coming to gym for other exercises (endurance training, cardiovascular training)

Ages: 19 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Bourbon TMS test (core strength) | 6 to 8 weeks
  The Bourbon Trunk Muscle Strength(TMS) test is an economical measure for assessment of dorsal, ventral and lateral trunk muscle chains.

SECONDARY OUTCOMES:
Stand-and-reach test (flexibility) | 6 to 8 weeks
  It is used for the measurement of spinal and pelvic flexibility. Excellent test-retest reliability has been reported for the stand-and-reach test with an ICC of 0.94.
20-m sprint test (speed) | 6 to 8 weeks
  Maximum effort sprints will be assessed from a stationary start to a distance of 20 meters to assess the speed of participant. Excellent test-retest reliability has been reported for the hand stopped 20-m sprint test with an intra-class correlation coefficient (ICC) of 0.90 variable
Jumping Sideways Test | 6 to 8 weeks
  The jumping sideways test evaluates motor coordination under time pressure. Excellent test-retest reliability has been reported for the jumping sideways test with an ICC of 0.89
Y Balance Test | 6 to 8 weeks
  The lower quarter Y balance test is a dynamic test that requires subjects to maintain single leg stance while reaching as far as possible with the contralateral leg in 3 different movement directions (i.e., anterior, posteromedial, posterolateral). Excellent test retest reliability has been reported for the Y balance test in all 3 movement directions with ICC values ranging between 0.89 and 0.93.

CONTACTS AND LOCATIONS:
Overall Officials: Raeed Mufti, MSPT-SPT, Principal Investigator — Riphah International University
Locations (1):
- Contours Gym Rehman Medical Institute, Peshawar, Khyberpakhtunkhuaw, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Imai A, Kaneoka K, Okubo Y, Shiina I, Tatsumura M, Izumi S, Shiraki H. Trunk muscle activity during lumbar stabilization exercises on both a stable and unstable surface. J Orthop Sports Phys Ther. 2010 Jun;40(6):369-75. doi: 10.2519/jospt.2010.3211. PMID 20511695
- [Background] Escamilla RF, Lewis C, Bell D, Bramblet G, Daffron J, Lambert S, Pecson A, Imamura R, Paulos L, Andrews JR. Core muscle activation during Swiss ball and traditional abdominal exercises. J Orthop Sports Phys Ther. 2010 May;40(5):265-76. doi: 10.2519/jospt.2010.3073. PMID 20436242
- [Background] Kim K-J. Effects of Core Muscle Strengthening Training on Flexibility, Muscular Strength and Driver Shot Performance in Female Professional Golfers. International Journal of Applied sports sciences. 2010;22(1).
- [Background] Kahle N, Tevald MA. Core muscle strengthening's improvement of balance performance in community-dwelling older adults: a pilot study. J Aging Phys Act. 2014 Jan;22(1):65-73. doi: 10.1123/japa.2012-0132. Epub 2013 Jan 23. PMID 23348043
- [Background] Okada T, Huxel KC, Nesser TW. Relationship between core stability, functional movement, and performance. J Strength Cond Res. 2011 Jan;25(1):252-61. doi: 10.1519/JSC.0b013e3181b22b3e. PMID 20179652
- [Background] Martuscello JM, Nuzzo JL, Ashley CD, Campbell BI, Orriola JJ, Mayer JM. Systematic review of core muscle activity during physical fitness exercises. J Strength Cond Res. 2013 Jun;27(6):1684-98. doi: 10.1519/JSC.0b013e318291b8da. PMID 23542879
- [Background] Uribe BP, Coburn JW, Brown LE, Judelson DA, Khamoui AV, Nguyen D. Muscle activation when performing the chest press and shoulder press on a stable bench vs. a Swiss ball. J Strength Cond Res. 2010 Apr;24(4):1028-33. doi: 10.1519/JSC.0b013e3181ca4fb8. PMID 20300023
- [Background] Kim MH, Oh JS. Effects of performing an abdominal hollowing exercise on trunk muscle activity during curl-up exercise on an unstable surface. J Phys Ther Sci. 2015 Feb;27(2):501-3. doi: 10.1589/jpts.27.501. Epub 2015 Feb 17. PMID 25729202
- [Background] Lago-Fuentes C, Rey E, Padron-Cabo A, Sal de Rellan-Guerra A, Fragueiro-Rodriguez A, Garcia-Nunez J. Effects of Core Strength Training Using Stable and Unstable Surfaces on Physical Fitness and Functional Performance in Professional Female Futsal Players. J Hum Kinet. 2018 Dec 31;65:213-224. doi: 10.2478/hukin-2018-0029. eCollection 2018 Dec. PMID 30687433
- [Background] Axel TA, Crussemeyer JA, Dean K, Young DE. Field Test Performance of Junior Competitive Surf Athletes following a Core Strength Training Program. Int J Exerc Sci. 2018 Jun 1;11(6):696-707. doi: 10.70252/XHXE2254. eCollection 2018. PMID 29997737
- [Background] Hsu SL, Oda H, Shirahata S, Watanabe M, Sasaki M. Effects of core strength training on core stability. J Phys Ther Sci. 2018 Aug;30(8):1014-1018. doi: 10.1589/jpts.30.1014. Epub 2018 Jul 24. PMID 30154592
- [Background] Thompson WR. Worldwide survey of fitness trends for 2018: the CREP edition. ACSM's Health & Fitness Journal. 2017;21(6):10-9.